CLINICAL TRIAL: NCT03571932
Title: Assessment of Family Planning and Immunization Service Integration in Liberia
Status: Completed | Type: Observational
Sponsor: Jhpiego (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); John Snow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00007524
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Contraception; Contraceptive Usage; Contraception Behavior; Infant, Newborn, Diseases
MeSH Terms: conditions — Contraception Behavior; Infant, Newborn, Diseases | interventions — Family Planning Services

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Facilities: Includes 18 health facilities
  Interventions: Behavioral: Family planning and immunization service integration
- Comparison facilities: Infludes 18 health facilities

INTERVENTIONS:
Behavioral: Family planning and immunization service integration — The approach involved integration of immunization and family planning services at health facilities. Vaccinators provided brief FP messages one-on-one to mothers and offered a referral for same-day, co-located FP services at the end of each routine immunization visit. For women coming directly for FP, if women had an infant with them, FP providers asked to see the child's health card, checked the return date for the next vaccination and reminded the mother of the date to return. For women without their child or the child health card with them, FP providers reinforced the importance of vaccination, and encouraged the mothers to bring their child for all their vaccines and complete the immunization schedule in a timely manner. A job aid, referral cards, and IEC materials were introduced to support the integration process.
  Groups: Intervention Facilities

SUMMARY:
This is a mixed methods process evaluation of a programmatic intervention to integrate family planning and immunization services at health facilities in Lofa and Grand Bassa counties in Liberia. MCSP used a longitudinal, pair-matched design to monitor the effect of integrating immunization and FP services on utilization of FP and routine immunization services. In Lofa and Grand Bassa counties, 36 facilities were pair-matched to intervention and comparison sites based on predetermined criteria. After approximately 9 months of implementation, MCSP conducted a qualitative study employing key informant interviews (KIIs) and focus group discussions (FGDs) at intervention and comparison sites, and with district-, county-, and national-level MOH supervisors and managers.

ELIGIBILITY:
Inclusion Criteria:

* 18 intervention facilities in Lofa and Grand Bassa counties
* 18 pair matched comparison facilities in Lofa and Grand Bassa counties

Exclusion Criteria:

* Facilities not included in the intervention or selected for pair matching

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 18 Intervention health facilities and 18 pair matched comparison health facilities in Grand Bassa and Lofa counties.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of modern family planning users | November 2016-July 2017
Number of Penta 1 doses administered | November 2016-July 2017
Number of Penta 3 doses administered | November 2016-July 2017

IPD SHARING:
Plan to Share IPD: No